CLINICAL TRIAL: NCT02610868
Title: A Phase 3, Long-Term, Open-Label and Single-Arm Study of MYOBLOC® in the Treatment of Troublesome Sialorrhea in Adult Subjects
Brief Title: Open-Label and Single-Arm Study of MYOBLOC® in the Treatment of Troublesome Sialorrhea in Adults
Acronym: OPTIMYST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SN-SIAL-351
Record Dates: First submitted 2015-11-02; First posted 2015-11-20 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2019-11

CONDITIONS: Sialorrhea
Keywords: Cerebral Palsy; ALS; Stroke; Neuroleptics
MeSH Terms: conditions — Sialorrhea; Cerebral Palsy; Stroke | interventions — rimabotulinumtoxinB

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MYOBLOC Injection (Experimental): After a screening period (up to 21 days), subjects who satisfy all eligibility criteria may receive single dose injections over the course of 1 year.
  Interventions: Drug: MYOBLOC

INTERVENTIONS:
Drug: MYOBLOC — After a screening period (up to 21 days), subjects who satisfy all eligibility criteria may receive single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments via injections into the submandibular and parotid glands. Subjects will undergo safety and effectiveness assessments at Weeks 4, 8, 13, 17, 26, 30, 39, 43, and 52, and telephone follow up will occur at Weeks 21, 34, and 47
  Other Names: rimabotulinumtoxinB; botulinum toxin type B

SUMMARY:
Multicenter, open-label, outpatient study of the safety and effectiveness of repeated doses of MYOBLOC over a 1-year duration in adult subjects with troublesome sialorrhea.

DETAILED DESCRIPTION:
Multicenter, open-label, outpatient study of the safety and effectiveness of repeated doses of MYOBLOC over a 1-year duration in adult subjects with troublesome sialorrhea. The primary goal is to determine the long-term safety and tolerability of MYOBLOC (administered intraglandularly as single total dose of 3,500 Units) treatments every 13 weeks over a maximum possible duration of 1 year in adult subjects with troublesome sialorrhea. The secondary goal is to assess the magnitude of therapeutic response of MYOBLOC (administered intraglandularly as a single total dose of 3,500 Units) using effectiveness assessments performed at intervals after treatments every 13 weeks over a maximum possible duration of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment for troublesome sialorrhea for at least 3 months that is occurring secondary to any disorder or related to any cause, including, but not limited to, Parkinson's Disease (PD), adult cerebral palsy, amyotrophic lateral sclerosis (ALS), stroke, traumatic brain injury, oral cancer, and side effects of other medications.
* Able to read and provide written informed consent before enrollment into the study, or the subject's caregiver (Legally Authorized Representative) can provide written informed consent.
* Male or female, 18 to 85 years of age (inclusive).
* Minimum unstimulated salivary flow rate of 0.2 g/min at screening
* Minimum Investigator's Drooling Frequency and Severity Scale (DFSS) score of 4 at screening.
* Ability and availability to participate in the study for up to 1 year (ALS subjects: ability and availability to participate in the study for at least 6 months), based on overall health of the subject and disease prognosis

Exclusion Criteria:

* A moderate to high risk of aspiration will exclude participation in this study. Subjects whose risk of aspiration are judged by the Investigator to be satisfactorily controlled by placement of PEG tube or G-tube for nutritional support are eligible to participate.
* Respiratory forced vital capacity (FVC) of <20% of predicted
* Prior botulinum toxin type A or B treatment in the salivary gland(s) identified for treatment in this study within 24 weeks before screening. Prior botulinum toxin type A or B treatment into other anatomical regions not selected for treatment in this study is not exclusionary, but must have occurred at least 12 weeks before screening
* Subjects should be excluded if, in the Investigator's opinion, the subject failed to respond to previous treatment with botulinum toxin. Subjects should not receive nor have any plans for receiving any botulinum toxin treatment, other than the study drug (MYOBLOC), during the entire course of the study (from the point the informed consent is signed until subject's participation is complete).
* Concomitant use, or exposure within 5 half-lives of screening, of aminoglycoside antibiotics, curare-like agents, or other agents that interfere with neuromuscular function
* Prior salivary gland surgery
* Current treatment or treatment at any time during the study with Coumadin® (warfarin) or similar anti-coagulant medications. Anti-platelet medications are not specifically exclusionary
* Evidence of any clinically significant neurologic disease
* Pregnancy or lactation
* Anticipated or scheduled surgery during the study period. A PEG tube/G tube may be placed for nutritional support at any time during the study and will not exclude the subject from continued study participation.
* Major surgery (requiring general anesthesia, except PEG tube/G tube placement ) within the previous 6 months before screening.
* Current infection at the sialorrhea treatment injection site(s)
* History of drug or alcohol abuse currently or within the previous 6 months
* Participation in another clinical drug, device, or biological agent study within 30 days of screening or while participating in this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Najeebah Abdul-Musawir, MD,MBA, Study Director — Supernus Pharmaceuticals, Inc.
Locations (34):
- United States (25):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Loma Linda, California
  - Los Angeles, California
  - Aurora, Colorado
  - Atlantis, Florida
  - Boca Raton, Florida
  - Orlando, Florida
  - Port Charlotte, Florida
  - Atlanta, Georgia
  - Kansas City, Kansas
  - Overland Park, Kansas
  - Elkridge, Maryland
  - Farmington Hills, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Edison, New Jersey
  - Centerville, Ohio
  - Tulsa, Oklahoma
  - Greenville, South Carolina
  - Cordova, Tennessee
  - San Antonio, Texas
  - Kirkland, Washington
  - Spokane, Washington
  - Tacoma, Washington
- Grodno, Belarus
- Ukraine (8):
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Kharkiv
  - Lviv
  - Odesa
  - Rivne
  - Uzhhorod
  - Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pahwa R, Molho E, Lew M, Dashtipour K, Gil RA, Revilla FJ, Clinch T, Qin P, Isaacson SH; OPen Label Trial of Intraglandular MYobloc injections for Sialorrhea Treatment (OPTIMYST) study group. Long-Term Safety and Efficacy of Repeated Cycles of RimabotulinumtoxinB in the Treatment of Chronic Sialorrhea: Results of the OPTIMYST Trial. Neurol Ther. 2025 Aug;14(4):1553-1567. doi: 10.1007/s40120-025-00777-z. Epub 2025 Jun 11. PMID 40498248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per protocol participants were only required to complete two treatment sessions with a maximum of 4 treatment sessions allowed.
Pre-assignment Details: All subjects received 3500 U doses except for 13 subjects who had decreased doses at Treatment Session 2 and/or 3 (2500 U to 3000 U).
Groups:
- MYOBLOC: 3500U: After a screening period (up to 21 days), subjects who satisfy all eligibility criteria may receive single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments.
Period: MYOBLOC: Treatment Session 1
Arm/Group | MYOBLOC: 3500U
Started | 187
Completed | 180
Not Completed | 7
Period: MYOBLOC: Treatment Session 2
Arm/Group | MYOBLOC: 3500U
Started | 177
Completed | 165
Not Completed | 12
Period: MYOBLOC: Treatment Session 3
Arm/Group | MYOBLOC: 3500U
Started | 50
Completed | 43
Not Completed | 7
Period: MYOBLOC: Treatment Session 4
Arm/Group | MYOBLOC: 3500U
Started | 24
Completed | 22
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Eligible subjects included male or females aged 18 to 85 years who are seeking treatment for troublesome sialorrhea for at least 3 months before screening.
Groups:
- MYOBLOC: MYOBLOC: After a screening period (up to 21 days), subjects who satisfy all eligibility criteria may receive single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments via injections into the submandibular and parotid glands. Subjects will undergo safety and effectiveness assessments at Weeks 4, 8, 13 for Treatment Session 1; Weeks 4, 13 for Treatment Sessions 2-4.
  All subjects received 3500 U doses except for 13 subjects who had decreased doses at Treatment Session 2 and/or 3 (2500 U to 3000 U).
Arm/Group | MYOBLOC
Number analyzed (Participants) | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 85
  >=65 years | 102
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 175
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 68
  Ukraine | 80
  Belarus | 39
Unstimulated Salivary Flow Rate (USFR) [Mean (Standard Deviation); unit: g/minute] | 0.6322 (0.4918)
Clinical Global Impression of Severity (CGI-S) [Mean (Standard Deviation); unit: units on a scale (1-7)] | 4.4 (0.94)
Patient Global Impression of Severity (PGI-S) [Mean (Standard Deviation); unit: units on a scale (1-7)] | 5.3 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence, Seriousness, Severity, and Causality Assessment of Treatment Emergent Adverse Events (TEAE)
Description: TEAEs Related to Study Medication include TEAEs classified as Possibly, Probably and Definitely Related.
  Treatment Session (TS)
Time Frame: Visits at Weeks 4 and 13 combined for each TS; including Visit at Week 8 for TS1
Population: Per protocol participants were only required to complete two treatment sessions with a maximum of 4 treatment sessions allowed.
  All subjects received 3500 U doses except for 13 subjects who had decreased doses at Treatment Session 2 and/or 3 (2500 U or 3000 U).
Measure: Number; unit: participants
Groups:
- Treatment Session 1; Treatment Session 2; Treatment Session 3; Treatment Session 4: Subjects received single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments. Subjects will undergo safety and effectiveness assessments.
Arm/Group | Treatment Session 1 | Treatment Session 2 | Treatment Session 3 | Treatment Session 4
Number analyzed (Participants) | 187 | 177 | 50 | 24
participants
  Serious TEAEs | 7 | 14 | 3 | 2
  Severe TEAEs | 5 | 8 | 2 | 2
  TEAEs Related to Study Medication | 42 | 26 | 4 | 2

2. Primary Outcome: Occurrence of Adverse Events of Special Interest (AESI)
Description: Treatment Session (TS)
  AESI includes: Aspiration, Aspirational pneumonia, Choking and Dysphagia.
Time Frame: Visits at Weeks 4 and 13 combined for each TS; including Visit at Week 8 for TS1
Population: Per protocol participants were only required to complete two treatment sessions with a maximum of 4 treatment sessions allowed.
  All subjects received 3500 U doses except for 13 subjects who had decreased doses at Treatment Session 2 and/or 3 (2500 U to 3000 U).
Measure: Number; unit: participants
Arm/Group | Treatment Session 1 | Treatment Session 2 | Treatment Session 3 | Treatment Session 4
Number analyzed (Participants) | 187 | 177 | 50 | 24
participants
  Aspiration | 0 | 1 | 0 | 0
  Aspirational pneumonia | 0 | 1 | 0 | 0
  Choking | 0 | 0 | 0 | 0
  Dysphagia | 4 | 0 | 0 | 0

3. Primary Outcome: Columbia Suicide Rating Scale (C-SSRS): Suicidal Ideation, Behavior Scores and Intensity Scores
Description: Participants Analyzed does not match the Participant Flow because one participant discontinued prior to the first post-injection visit.
  Per protocol participants were only required to complete two treatment sessions with a maximum of 4 treatment sessions allowed.
  All subjects received 3500 U doses except for 13 subjects who had decreased doses at Treatment Session 2 and/or 3 (2500 U to 3000 U).
Time Frame: Baseline (Day 1) of each TS to the following: TS1 Visits at Weeks 4, 8, 13; TS2-4 Visits at Weeks 4, 13
Measure: Number; unit: participants
Groups:
- Treatment Session 1: Week 4; Treatment Session 1: Week 8; Treatment Session 1: Week 13: Subjects received single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments. Subjects will undergo safety and effectiveness assessments for Treatment Session 1 at Weeks 4, 8, 13.
- Treatment Session 2: Week 4; Treatment Session 2: Week 13: Subjects received single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments. Subjects will undergo safety and effectiveness assessments for Treatment Session 2 at Weeks 4 and 13.
- Treatment Session 3: Week 4; Treatment Session 3: Week 13: Subjects received single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments. Subjects will undergo safety and effectiveness assessments for Treatment Session 3 at Weeks 4 and 13.
- Treatment Session 4: Week 4; Treatment Session 4: Week 13: Subjects received single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments. Subjects will undergo safety and effectiveness assessments for Treatment Session 4 at Weeks 4 and 13.
Arm/Group | Treatment Session 1: Week 4 | Treatment Session 1: Week 8 | Treatment Session 1: Week 13 | Treatment Session 2: Week 4 | Treatment Session 2: Week 13 | Treatment Session 3: Week 4 | Treatment Session 3: Week 13 | Treatment Session 4: Week 4 | Treatment Session 4: Week 13
Number analyzed (Participants) | 186 | 183 | 181 | 175 | 166 | 49 | 45 | 24 | 23
participants
  Suicidal Ideation | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Suicidal Behavior | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Occurrence of Dental Adverse Events
Description: Treatment Session (TS)
Time Frame: Visits at Weeks 4 and 13 combined for each TS; including Visit at Week 8 for TS1
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Treatment Session 1 | Treatment Session 2 | Treatment Session 3 | Treatment Session 4
Number analyzed (Participants) | 187 | 177 | 50 | 24
participants | 27 | 23 | 8 | 2

5. Secondary Outcome: Change From Baseline in Unstimulated Salivary Flow Rate (USFR): Treatment Sessions 1-4
Description: For Treatment Sessions 2-4, the change from baseline is calculated using the Week 13 value from the previous Treatment Session as the new baseline. Week 8 was only assessed in Treatment Session 1.
  Treatment Session (TS)
  Participants Analyzed does not match the Participant Flow because patient data was not always captured for each endpoint at every visit.
Time Frame: Baseline (Day 1) of each TS to the following: TS1 Visits at Weeks 4, 8, 13; TS2-4 Visits at Weeks 4, 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/minute
Arm/Group | Treatment Session 1: Week 4 | Treatment Session 1: Week 8 | Treatment Session 1: Week 13 | Treatment Session 2: Week 4 | Treatment Session 2: Week 13 | Treatment Session 3: Week 4 | Treatment Session 3: Week 13 | Treatment Session 4: Week 4 | Treatment Session 4: Week 13
Number analyzed (Participants) | 185 | 183 | 181 | 174 | 166 | 49 | 45 | 24 | 23
g/minute | -0.3424 (0.3685) | -0.2771 (0.3144) | -0.1357 (0.2888) | -0.2272 (0.2668) | -0.0560 (0.2067) | -0.1797 (0.1975) | -0.0547 (0.2269) | -0.1592 (0.2305) | -0.0335 (0.1378)
Statistical Analysis 1: Comparison: Treatment Session 1: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Treatment Session 1: Week 8; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: Treatment Session 1: Week 13; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: Treatment Session 2: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 5: Comparison: Treatment Session 2: Week 13; Test type: Superiority; p = 0.0006, ANCOVA
Statistical Analysis 6: Comparison: Treatment Session 3: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 7: Comparison: Treatment Session 3: Week 13; Test type: Superiority; p = 0.1131, ANCOVA
Statistical Analysis 8: Comparison: Treatment Session 4: Week 4; Test type: Superiority; p = 0.0026, ANCOVA
Statistical Analysis 9: Comparison: Treatment Session 4: Week 13; Test type: Superiority; p = 0.2569, ANCOVA

6. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S)
Description: CGI-S will be used to record the severity of illness (sialorrhea) on a 7-point scale ranging from a score of 1, "normal" to a score of 7, "among the most extremely ill patients".
  Treatment Session (TS)
  Participants Analyzed does not match the Participant Flow because participant discontinued prior to the first post-injection visit.
Time Frame: Baseline (Day 1) of each TS to the following: TS1 Visits at Weeks 4, 8, 13; TS2-4 Visits at Weeks 4, 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Session 1: Week 4 | Treatment Session 1: Week 8 | Treatment Session 1: Week 13 | Treatment Session 2: Week 4 | Treatment Session 2: Week 13 | Treatment Session 3: Week 4 | Treatment Session 3: Week 13 | Treatment Session 4: Week 4 | Treatment Session 4: Week 13
Number analyzed (Participants) | 186 | 183 | 181 | 175 | 167 | 49 | 45 | 24 | 23
units on a scale | -1.7 (1.26) | -1.5 (1.22) | -0.9 (1.03) | -0.8 (1.12) | -0.1 (0.99) | -0.9 (1.13) | -0.2 (0.90) | -0.9 (0.95) | -0.3 (1.02)
Statistical Analysis 1: Comparison: Treatment Session 1: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Treatment Session 1: Week 8; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: Treatment Session 1: Week 13; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: Treatment Session 2: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 5: Comparison: Treatment Session 2: Week 13; Test type: Superiority; p = 0.3130, ANCOVA
Statistical Analysis 6: Comparison: Treatment Session 3: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 7: Comparison: Treatment Session 3: Week 13; Test type: Superiority; p = 0.1054, ANCOVA
Statistical Analysis 8: Comparison: Treatment Session 4: Week 4; Test type: Superiority; p = 0.0002, ANCOVA
Statistical Analysis 9: Comparison: Treatment Session 4: Week 13; Test type: Superiority; p = 0.1663, ANCOVA

7. Secondary Outcome: Clinical Global Impression of Change (CGI-C)
Description: CGI-C will be used to record change or improvement of illness (sialorrhea) on a 7-point scale ranging from a score of 1, "very much improved" to a score of 7, "very much worse".
  Participants Analyzed does not match the Participant Flow because participant discontinued prior to the first post-injection visit.
  Treatment Session (TS)
Time Frame: TS1 Visits at Weeks 4, 8, 13; TS2-4 Visits at Weeks 4, 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Session 1: Week 4 | Treatment Session 1: Week 8 | Treatment Session 1: Week 13 | Treatment Session 2: Week 4 | Treatment Session 2: Week 13 | Treatment Session 3: Week 4 | Treatment Session 3: Week 13 | Treatment Session 4: Week 4 | Treatment Session 4: Week 13
Number analyzed (Participants) | 186 | 183 | 181 | 175 | 167 | 49 | 45 | 24 | 23
units on a scale | 2.3 (0.94) | 2.4 (1.07) | 3.0 (1.16) | 2.4 (1.04) | 3.1 (1.34) | 2.4 (0.94) | 3.0 (1.06) | 2.5 (0.93) | 2.8 (0.94)

8. Secondary Outcome: Change From Baseline in Drooling Frequency and Severity Scale Performed by Trained Assessor (DFSS-I)
Description: The DFSS will be used to assess the frequency and severity of drooling on a 5-point scale ranging from a score of 1, dry never drools to a score of 5, profuse clothing hands tray objects become wet. Drooling frequency will be assessed on a 4-point scale ranging from a score of 1, never drools to a score of 4, constantly drools.
  Treatment Session (TS)
  Participants Analyzed does not match the Participant Flow because participant discontinued prior to the first post-injection visit.
  The severity score and frequency score are summed together to create the DFSS total score (range 2-9). A decrease from baseline indicates improvement.
Time Frame: Baseline (Day 1) of each TS to the following: TS1 Visits at Weeks 4, 8, 13; TS2-4 Visits at Weeks 4, 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Session 1: Week 4 | Treatment Session 1: Week 8 | Treatment Session 1: Week 13 | Treatment Session 2: Week 4 | Treatment Session 2: Week 13 | Treatment Session 3: Week 4 | Treatment Session 3: Week 13 | Treatment Session 4: Week 4 | Treatment Session 4: Week 13
Number analyzed (Participants) | 186 | 783 | 181 | 175 | 167 | 49 | 45 | 24 | 23
units on a scale | -2.3 (1.53) | -2.0 (1.52) | -1.2 (1.37) | -1.2 (1.52) | -0.2 (1.30) | -1.1 (1.36) | 0.0 (1.33) | -1.5 (1.44) | -0.3 (0.71)
Statistical Analysis 1: Comparison: Treatment Session 1: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Treatment Session 1: Week 8; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: Treatment Session 1: Week 13; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: Treatment Session 2: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 5: Comparison: Treatment Session 2: Week 13; Test type: Superiority; p = 0.1100, ANCOVA
Statistical Analysis 6: Comparison: Treatment Session 3: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 7: Comparison: Treatment Session 3: Week 13; Test type: Superiority; p = 1.0000, ANCOVA
Statistical Analysis 8: Comparison: Treatment Session 4: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 9: Comparison: Treatment Session 4: Week 13; Test type: Superiority; p = 0.0290, ANCOVA

9. Secondary Outcome: Change From Baseline in Drooling Frequency and Severity Scale Performed by Subject (DFSS-S)
Description: The DFSS will be used to assess the frequency and severity of drooling on a 5-point scale ranging from a score of 1, dry never drools to a score of 5, profuse clothing hands tray objects become wet. Drooling frequency will be assessed on a 4-point scale ranging from a score of 1, never drools to a score of 4, constantly drools.
  Treatment Session (TS)
  Participants Analyzed does not match the Participant Flow because patient data was not always captured for each endpoint at every visit.
  The severity score and frequency score are summed together to create the DFSS total score (range 2 -9). A decrease from baseline indicates improvement.
Time Frame: Baseline (Day 1) of each TS to the following: TS1 Visits at Weeks 4, 8, 13; TS2-4 Visits at Weeks 4, 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Session 1: Week 4 | Treatment Session 1: Week 8 | Treatment Session 1: Week 13 | Treatment Session 2: Week 4 | Treatment Session 2: Week 13 | Treatment Session 3: Week 4 | Treatment Session 3: Week 13 | Treatment Session 4: Week 4 | Treatment Session 4: Week 13
Number analyzed (Participants) | 184 | 182 | 177 | 170 | 162 | 48 | 43 | 23 | 22
units on a scale | -1.4 (1.35) | -1.7 (1.58) | -1.0 (1.49) | -0.7 (0.90) | -0.3 (0.98) | -0.4 (0.64) | 0.0 (1.00) | -0.4 (1.03) | -0.2 (1.37)
Statistical Analysis 1: Comparison: Treatment Session 1: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Treatment Session 1: Week 8; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: Treatment Session 1: Week 13; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: Treatment Session 2: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 5: Comparison: Treatment Session 2: Week 13; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 6: Comparison: Treatment Session 3: Week 4; Test type: Superiority; p = 0.0003, ANCOVA
Statistical Analysis 7: Comparison: Treatment Session 3: Week 13; Test type: Superiority; p = 0.9016, ANCOVA
Statistical Analysis 8: Comparison: Treatment Session 4: Week 4; Test type: Superiority; p = 0.0753, ANCOVA
Statistical Analysis 9: Comparison: Treatment Session 4: Week 13; Test type: Superiority; p = 0.4992, ANCOVA

10. Secondary Outcome: Change From Baseline in Patient Global Impression of Severity (PGI-S)
Description: The PGI-S scale will be used by the subject to rate the severity of his/her illness (sialorrhea) on an 7-point scale ranging from a score of 1, "normal" to a score of 7, "among the most extremely ill".
  Treatment Session (TS)
  Participants Analyzed does not match the Participant Flow because participant discontinued prior to the first post-injection visit.
Time Frame: Baseline (Day 1) of each TS to the following: TS1 Visits at Weeks 4, 8, 13; TS2-4 Visits at Weeks 4, 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Session 1: Week 4 | Treatment Session 1: Week 8 | Treatment Session 1: Week 13 | Treatment Session 2: Week 4 | Treatment Session 2: Week 13 | Treatment Session 3: Week 4 | Treatment Session 3: Week 13 | Treatment Session 4: Week 4 | Treatment Session 4: Week 13
Number analyzed (Participants) | 186 | 183 | 181 | 174 | 167 | 49 | 45 | 24 | 23
units on a scale | -1.59 (1.548) | -1.41 (1.461) | -0.80 (1.364) | -0.78 (1.303) | -0.07 (1.245) | -0.94 (1.248) | 0.04 (1.242) | -1.38 (1.279) | -0.26 (1.251)
Statistical Analysis 1: Comparison: Treatment Session 1: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Treatment Session 1: Week 8; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: Treatment Session 1: Week 13; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: Treatment Session 2: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 5: Comparison: Treatment Session 2: Week 13; Test type: Superiority; p = 0.4567, ANCOVA
Statistical Analysis 6: Comparison: Treatment Session 3: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 7: Comparison: Treatment Session 3: Week 13; Test type: Superiority; p = 0.8115, ANCOVA
Statistical Analysis 8: Comparison: Treatment Session 4: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 9: Comparison: Treatment Session 4: Week 13; Test type: Superiority; p = 0.3282, ANCOVA

11. Secondary Outcome: Patient Global Impression of Change (PGI-C)
Description: The PGI-C scale will be used by the subject to rate the change in symptoms of his/her illness (sialorrhea) on an 7-point scale ranging from a score of 1, "very much improved" to a score of 7, "very much worse".
  Treatment Session (TS)
  Participants Analyzed does not match the Participant Flow because participant discontinued prior to the first post-injection visit.
Time Frame: TS1 Visits at Weeks 4, 8, 13; TS2-4 Visits at Weeks 4, 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Session 1: Week 4 | Treatment Session 1: Week 8 | Treatment Session 1: Week 13 | Treatment Session 2: Week 4 | Treatment Session 2: Week 13 | Treatment Session 3: Week 4 | Treatment Session 3: Week 13 | Treatment Session 4: Week 4 | Treatment Session 4: Week 13
Number analyzed (Participants) | 186 | 183 | 181 | 174 | 167 | 49 | 45 | 24 | 23
units on a scale | 2.5 (1.07) | 2.7 (1.08) | 3.0 (1.13) | 2.6 (1.06) | 3.2 (1.28) | 2.7 (0.95) | 3.2 (1.10) | 2.5 (0.72) | 3.4 (0.72)

12. Secondary Outcome: Change From Baseline in Drooling Impact Score (DIS)
Description: The DIS is a 10-item questionnaire with each item rated by the subject to evaluate the impact of sialorrhea on daily activities (e.g., speech, social activities).
  Treatment Session (TS)
  Participants Analyzed does not match the Participant Flow because patient data was not always captured for each endpoint at every visit.
  Subject is requested to compare their current status to their last study visit using a 4-point scale ranging from a score of 1, not at all to a score of 4, very much. The DIS total score ranges from 10 to 40. A negative change from baseline indicates a positive clinical outcome.
Time Frame: Baseline (Day 1) of each TS to the following: TS1 Visits at Weeks 4, 8, 13; TS2-4 Visits at Weeks 4, 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Session 1: Week 4 | Treatment Session 1: Week 8 | Treatment Session 1: Week 13 | Treatment Session 2: Week 4 | Treatment Session 2: Week 13 | Treatment Session 3: Week 4 | Treatment Session 3: Week 13 | Treatment Session 4: Week 4 | Treatment Session 4: Week 13
Number analyzed (Participants) | 185 | 183 | 181 | 175 | 167 | 49 | 45 | 24 | 23
units on a scale | -5.2 (5.33) | -5.4 (5.16) | -3.4 (4.97) | -2.5 (4.17) | 0.3 (3.94) | -2.8 (3.39) | -0.1 (2.11) | -3.6 (3.10) | -0.5 (2.57)
Statistical Analysis 1: Comparison: Treatment Session 1: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Treatment Session 1: Week 8; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: Treatment Session 1: Week 13; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: Treatment Session 2: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 5: Comparison: Treatment Session 2: Week 13; Test type: Superiority; p = 0.3786, ANCOVA
Statistical Analysis 6: Comparison: Treatment Session 3: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 7: Comparison: Treatment Session 3: Week 13; Test type: Superiority; p = 0.7787, ANCOVA
Statistical Analysis 8: Comparison: Treatment Session 4: Week 4; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 9: Comparison: Treatment Session 4: Week 13; Test type: Superiority; p = 0.3825, ANCOVA

ADVERSE EVENTS:
Time Frame: through study completion, up to 1 year
Description: Systematic Assessment: Office visits were conducted on Weeks 4, 8, 13 for Treatment Session 1 and Weeks 4 and 13 for Treatment Sessions 2, 3, 4.
Groups:
- MYOBLOC: Treatment Session 1: After a screening period (up to 21 days), subjects who satisfy all eligibility criteria may receive single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments. Subjects will undergo safety and effectiveness assessments for Treatment Session 1 at Weeks 4, 8, 13.
  All subjects received 3500 U doses except for 13 subjects who had decreased doses at Treatment Session 2 and/or 3 (2500 U to 3000 U).
- MYOBLOC: Treatment Session 2: After a screening period (up to 21 days), subjects who satisfy all eligibility criteria may receive single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments. Subjects will undergo safety and effectiveness assessments for Treatment Session 2 at Weeks 4 and 13.
  All subjects received 3500 U doses except for 13 subjects who had decreased doses at Treatment Session 2 and/or 3 (2500 U to 3000 U).
- MYOBLOC: Treatment Session 3: After a screening period (up to 21 days), subjects who satisfy all eligibility criteria may receive single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments. Subjects will undergo safety and effectiveness assessments for Treatment Session 3 at Weeks 4 and 13.
  All subjects received 3500 U doses except for 13 subjects who had decreased doses at Treatment Session 2 and/or 3 (2500 U to 3000 U).
- MYOBLOC: Treatment Session 4: After a screening period (up to 21 days), subjects who satisfy all eligibility criteria may receive single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments. Subjects will undergo safety and effectiveness assessments for Treatment Session 4 at Weeks 4 and 13.
  All subjects received 3500 U doses except for 13 subjects who had decreased doses at Treatment Session 2 and/or 3 (2500 U to 3000 U).
- ALL MYOBLOC: Treatment Sessions 1-4: After a screening period (up to 21 days), subjects who satisfy all eligibility criteria may receive single dose injections of 3,500 Units of MYOBLOC every 13 weeks (±2 weeks) for a total of 4 treatments. Subjects will undergo safety and effectiveness assessments at Weeks 4, 8, 13 for Treatment Session 1, Weeks 4 and 13 for Treatment Sessions 2-4.
  All subjects received 3500 U doses except for 13 subjects who had decreased doses at Treatment Session 2 and/or 3 (2500 U to 3000 U).
Arm/Group | MYOBLOC: Treatment Session 1 | MYOBLOC: Treatment Session 2 | MYOBLOC: Treatment Session 3 | MYOBLOC: Treatment Session 4 | ALL MYOBLOC: Treatment Sessions 1-4
All-Cause Mortality (participants affected / at risk) | 1/187 | 4/177 | 2/50 | 1/24 | 8/187
Serious Adverse Events (participants affected / at risk) | 9/187 | 18/177 | 4/50 | 2/24 | 33/187
Other Adverse Events (participants affected / at risk) | 44/187 | 34/177 | 7/50 | 4/24 | 73/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MYOBLOC: Treatment Session 1 (N=187) | MYOBLOC: Treatment Session 2 (N=177) | MYOBLOC: Treatment Session 3 (N=50) | MYOBLOC: Treatment Session 4 (N=24) | ALL MYOBLOC: Treatment Sessions 1-4 (N=187)
Angina pectoris (Cardiac disorders) | 2 | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Post procedural compication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 2
Multiple system atrophy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 2 | 1 | 1 | 4 — Captured ALS subjects progression of disease.
Freezing phenomenon (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 1 | 0 | 3
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MYOBLOC: Treatment Session 1 (N=187) | MYOBLOC: Treatment Session 2 (N=177) | MYOBLOC: Treatment Session 3 (N=50) | MYOBLOC: Treatment Session 4 (N=24) | ALL MYOBLOC: Treatment Sessions 1-4 (N=187)
Dental caries (Gastrointestinal disorders) | 13 | 17 | 6 | 2 | 32
Dry mouth (Gastrointestinal disorders) | 29 | 10 | 1 | 0 | 33
Amyotrophic lateral sclerosis (Nervous system disorders) | 2 | 7 | 0 | 2 | 8 — Captured ALS subjects progression of disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-07-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT02610868/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT02610868/SAP_001.pdf